CLINICAL TRIAL: NCT02715778
Title: Translational Investigation of Gestational Environment on Neurobehavioral Function in Children
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Lee S. Cohen, MD, Professor of Psychiatry, Massachusetts General Hospital
Other Study IDs: 2015P001326
Record Dates: First submitted 2016-02-05; First posted 2016-03-22 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adult Participants
- Child Participants

SUMMARY:
Although the last decade has brought major advances with respect to our knowledge of certain risks associated with fetal exposure to psychiatric medications, critical information regarding the long-term neurobehavioral impact of fetal exposure is lacking. With a prevalence rate of selective serotonin reuptake inhibitor (SSRI) use across pregnancy in Western countries noted to be as high as 5-8%, this study aims to close the gap in knowledge regarding long-term neurobehavioral sequelae of in utero exposure to this class of antidepressants. Importantly, the assessment of the impact of antenatal psychotropic medication use must be conducted with an appreciation of the potential direct and indirect effects of maternal psychiatric illness during pregnancy and throughout childhood. The outcomes of this study will help to inform the care of reproductive age women treated with psychiatric medications as they, along with the clinicians prescribing for them, weigh the relative risks of using these agents during pregnancy.

DETAILED DESCRIPTION:
Neuropsychological evaluation of older children than previously studied with histories of fetal exposure to antidepressants and maternal depression during pregnancy is needed and may inform whether a signal for neural disruption exists following fetal selective serotonin reuptake inhibitor (SSRI) exposure. Identification of genetic factors which may afford resilience or particular vulnerability to fetal exposure to antidepressants is a logical component of this translational initiative designed to answer the proposed research question.

Because of the hypothesis that prenatal exposure to gamma-aminobutyric acid (GABA)-based drugs has the influence excitatory/inhibitory balance and to shift critical periods, there is reason to believe that some aspects of brain development may also be altered. To this end, this project aims to "scan" a variety of brain functions that include memory, attention, and executive functions; in addition, it will also examine the extent to which face and speech processing are altered in the target sample.

This study will assess older children ages 6-17 with histories of fetal exposure to antidepressants and/or maternal depression during pregnancy. It will evaluate child behavior based on maternal report and utilize neuropsychological evaluation to inform whether a signal for neural disruption exists following fetal SSRI or depression exposure. The neuropsychological assessments will be paired with an analysis of genetic factors which may afford resilience or particular vulnerability to fetal exposure to antidepressants.

This study leverages unique patient resources with respect to children of mothers with well documented histories of SSRI exposure who have been prospectively followed across pregnancy. The multidisciplinary collaboration between the lead investigator, Dr. Lee S. Cohen of the Center for Women's Mental Health (CWMH), and the Laboratories of Cognitive Neuroscience, Boston Children's Hospital (Dr. Charles Nelson), the Department of Molecular and Cellular Biology, and the Psychiatric and Neurodevelopmental Genetics Unit at Massachusetts General Hospital (Dr. Jordan Smoller) is a remarkable opportunity to better understand the effects of maternal antidepressant exposure during pregnancy on neuropsychological development of children.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal subjects:

   * have a child between 6-17 years of age
   * had a history of major depressive disorder (MDD) at the time of their pregnancy of the above child
   * are at least 18 years of age
2. Child subjects:

   * are between 6-17 years of age
   * are the children of women who fit the eligibility criteria described above and have consented to participate in the study
   * are able to provide informed assent and a parent or guardian is able and willing to provide informed consent

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will be composed of two components: a maternal assessment based at Massachusetts General Hospital (MGH) and a child evaluation based at Boston Children's Hospital. Mother and child pairs may elect to complete both components of the study. If either participant does not want the child to take part in the research, the maternal component may be completed alone. Similarly, the child may enroll in the research study without the enrollment of the mother with parental consent.
  Women who are interested and eligible for the study may choose to complete the study in-person at MGH or to be evaluated remotely by a phone interview and set of online surveys. All child subjects must participate in an in-person visit at Boston Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
neuropsychological functioning as assessed by CANTAB research battery | cross-sectional assessment at baseline (at 6-17 years of age, depending on subject's age at time of visit)
  Further information on CANTAB available at: http://www.cambridgecognition.com/academic/crs

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Cohen, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts